CLINICAL TRIAL: NCT04554810
Title: Improving Syrian Refugees' Knowledge of Medications and Adherence Following a Randomized Control Trial Assessing the Effect of a Medication Management Review Service
Brief Title: Pharmacists Improving Refugees' Adherence and Knowledge of Their Chronic Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Iman Basheti (Other)
Responsible Party: Sponsor-Investigator, Prof. Iman Basheti, Professor in Clinical Pharmacy, Applied Science Private University
Organization: Applied Science Private University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOH-REC-160079
Record Dates: First submitted 2020-09-08; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Diabetes; Hypertension; Dyslipidemias; Cardiac Disease; Asthma
Keywords: Refugees; Medication management review; Adherence; Pharmaceutical care; chronic medication; Jordan; Universal health coverage; Sustainable development goal
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Dyslipidemias; Heart Diseases; Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Intervention group participants are the refugees who received the medication management review service and pharmacist's counselling. They have been assessed at baseline and at follow-up after 3 months) home visits.
  Interventions: Other: Medication Management Service
- Control group (No Intervention): Control group participants are the refugees who did not received the medication management review service and no pharmacist's counselling wsa provided to them during the study period. They have been assessed at baseline and at follow-up (after 3 months) home visits.

INTERVENTIONS:
Other: Medication Management Service — Medication review was delivered to the Syrian refugees by accredited pharmacists at the baseline visit. This followed by identifying the treatment-related problems (TRP) by the clinical pharmacist, and correction of the approved TRPs by the corresponding physicians and finally convey these changes in medications to the patients. In addition, counselling and education were delivered to the refugees' patients in the base line visit.
  Arms: Intervention group

SUMMARY:
This study is a randomized, controlled, single-blinded clinical study which conducted over six months (May to October 2016) in different Jordanian cities, where most of Syrian refugees reside. The primary aim of this study was to assess refugees' adherence and knowledge of their chronic medications, and impact of the medication management review (MMR) service delivered by a clinical pharmacist on their adherence and knowledge of their chronic medications three months following delivering the service.

An informed consent form was signed by all participants who accepted to participate (n=106). Participants were then randomized into intervention and control groups. The first group would have received the medication management review service during the study period, while the to the other group directly after the study was completed (after three months' time). Two validated questionnaire were used in the study for assessment; adherence to medications questionnaire and Knowledge about chronic medications questionnaire. These questionnaire were filled by tha patients at baseline and follow up home visits.

DETAILED DESCRIPTION:
This study was a randomized interventional clinical study, conducted over six months (May to October 2016) in different Jordanian cities, where most of Syrian refugees reside. Clinics which are specialized for Syrian refugees were approached by the clinical pharmacist (researcher) in order to meet Syrian refugees, recruit eligible participants and arrange for their first home visits. An informed consent form was signed by all participants who accepted to participate. Participants were then randomized into intervention and control groups using a predetermined list obtained by the computer randomization program (www.randomizer.org). The study was single - blinded, hence, participants were not informed of the group they were randomized into, but they were informed that they would have been in either of two study groups. The first group would have received the medication management review (MMR) service during the study period, while the to the other group directly after the study was completed (after three months' time). Appointments were arranged at the physicians' clinics for all participants to be visited by the clinical pharmacist at their homes. At the baseline home visit, the clinical pharmacist documented participants' demographics, acute and chronic medical problems, history of present diseases, past medical history, lifestyle, family history, allergies, vital signs, physical examination information, diagnostic test data, lab results, current medications and issues related to the short and long term management of the patient .

The MMR service was completed following verification of collected baseline data. The home visits were planned not to exceed one hour. During these visits, self-completed questionnaires were completed by the participants, evaluating their adherence and knowledge about their chronic medications. The clinical pharmacist identified and documented the treatment-related problems (TRPs) for each patient in both groups at baseline. The physician was identified based on the participant's reported clinic and on participant's choice when more than one physician was visited by the participant. Following receipt of the letter, physicians addressed the recommendations and returned the letter to the pharmacist showing approved and rejected recommendations. Participants were called by the pharmacist to visit the physician and have the approved recommendations applied. Counselling and education were delivered to participants in the intervention group regarding their illnesses, knowledge of medications and adherence to their treatment. Three months post baseline, new appointments were arranged through a phone call by the clinical pharmacist, and all participants were revisited at home. Data needed to assess TRPs where recollected (as was done at baseline), plus the adherence and knowledge about chronic medications' questionnaires was completed for all participants. At the end of the study, control group participants received the MMR and pharmacist counselling service exactly as was delivered to the intervention group participants at baseline. For the purpose of data documentation and evaluation, the adherence to medication questionnaire and the knowledge about chronic medications were used. Data were coded then entered into the Statistical Package for Social Sciences (SPSS), version 20. Continuous variables were expressed as mean ± standard deviation . Differences within the same group were detected using paired sample t-test for continuous variables. Group differences (between the intervention and control groups) were detected using the independent sample t-test or Mann Whitney U-test (based on the normality of data following testing) for continuous variables. Categorical data were expressed as proportion (%) and analysed using Chi-square test. A probability value of < 0.05 was considered to be statistically significant for all analysis's tests.

ELIGIBILITY:
Inclusion Criteria:

* being Syrian refugee ≥ 18 years, living in Jordan for more than six months prior to study recruitment and intending to stay for the whole study period
* having one chronic condition at least or taking 5 or more medications or taking more than 12 doses of a medication per day

Exclusion Criteria:

* Patients with cognitive or sensory impairment that may prevent conducting the interview.
* Patients who are planning to travel within the next six months after the baseline home-visit
* Patients who are not capable of reading or writing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-05-10 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2016-01-30 (Actual)

PRIMARY OUTCOMES:
Adherence to medications scores | 3 months
  how often the patient during the last month forgot to take his/her medication/s, skipped it, stopped it when feeling better, stopped it when feeling worse or stopped it when they experienced a side effect. The measurement scale used in this questionnaire was scored at 0 (never), 1 (rarely), 2 (sometimes), 3 (often) and 4 (always). Hence, adherence was analysed as a continuous scale out of 32. Higher scores indicted lower adherence by the patient.
Knowledge about chronic medications scores | 3 months
  The questionnaire consisted of five questions related to patients' medications including 1- scientific medication name, 2- generic medication name, 3- how, 4- when, and 5- why was the patient taking each medication. The knowledge about medications was analysed as a continuous scale out of five. Higher scores indicated less knowledge about one's medication therapy.

CONTACTS AND LOCATIONS:
Overall Officials: I A Basheti, Study Director — Applied Science University, Amman, Jordan

REFERENCES:
- [Derived] Alalawneh M, Berardi A, Nuaimi N, Basheti IA. Improving Syrian refugees' knowledge of medications and adherence following a randomized control trial assessing the effect of a medication management review service. PLoS One. 2022 Oct 14;17(10):e0276304. doi: 10.1371/journal.pone.0276304. eCollection 2022. PMID 36240214